CLINICAL TRIAL: NCT07390916
Title: Expanded Use of Thermal Ablation (EXCEL Cohort) and Prophylactic Use of Two Probes (PRO Cohort) for Cervical Cancer Prevention in Women Living With HIV
Brief Title: Feasibility Study Comparing Use of One Or Two Probes for Thermal Ablation Among Cervical Cancer Screen Positive Women Living With HIV in C1001P-CS5 Rwanda
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Washington (Other); National Cancer Institute (NCI) (NIH); University of Cincinnati (Other); University of Rwanda (Other); Frontier Science & Technology Research Foundation, Inc. (Industry)
Responsible Party: Principal Investigator, Margaret M. Madeleine, PhD, Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1124082 (C1001P-CS5 Rwanda); UG1CA275402 (NIH); U24CA275417 (NIH)
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09

CONDITIONS: HIV (Human Immunodeficiency Virus); HPV; Cervical Precancer
Keywords: HIV; Cervical cancer screening; Treatment of Cervical Precancer; Thermal ablation; Human papillomavirus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Uterine Cervical Dysplasia

STUDY DESIGN:
Masking Description: Clinical Site staff involved in provision of clinical care, recruitment, or follow-up will be blinded to allocation until after visual inspection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (TA with 1 probe) (Experimental): Participants undergo a clinical exam, soft-brush endocervical and ectocervical biopsies, digital imaging, and visual assessment for TA, and if eligible undergo with 1 probe at month 0.
  Interventions: Procedure: Thermal ablation (TA) with 1 probe
- Group 2 (TA with 2 probes) (Experimental): Participants undergo a clinical exam, soft-brush endocervical and ectocervical biopsies, digital imaging, and visual assessment for TA, and if eligible undergo with 2 probes at month 0.
  Interventions: Procedure: Thermal ablation (TA) with 2 probes

INTERVENTIONS:
Procedure: Thermal ablation (TA) with 1 probe — Undergo TA with 1 probe
  Arms: Group 1 (TA with 1 probe)
Procedure: Thermal ablation (TA) with 2 probes — Undergo TA with 2 probes
  Arms: Group 2 (TA with 2 probes)

SUMMARY:
Cervical cancer disproportionately affects women in low- and middle-income countries (LMICs), particularly women living with HIV (WLWH) who have a 6-fold increased risk of cervical cancer compared to women in the general population. Thermal ablation (TA) is recommended by the World Health Organization (WHO) to treat cervical precancerous lesions, although its efficacy can be suboptimal in WLWH. This is even more important at a time when Rwanda has launched a National Cervical Cancer Screening Program (NCCSP) with human papillomavirus (HPV) testing and treatment, mainly using TA with unknown outcomes. Therefore, we will conduct a feasibility study (C1001P-CS5) among 300 Rwandan WLWH to provide evidence needed to launch a future effectiveness study. The proposed study will evaluate the feasibility, acceptability, and safety of a two-probe TA technique (endocervical and ectocervical probes) and whether this approach improves treatment outcomes among WLWH compared to one (ectocervical) probe. This innovation has the potential to significantly enhance cervical cancer prevention efforts in high-burden settings. It will also contribute towards achieving the 90-70-90 goals of the WHO strategy for accelerated elimination of cervical cancer as a public health problem by 2030. Rwanda hopes to achieve this goal early, in 2027 under Mission 2027.

DETAILED DESCRIPTION:
Participants will first undergo HPV testing or visual inspection with acetic acid at screening. Participants with positive screening results undergo a clinical exam comprising visual inspection with acetic acid, digital imaging, brush biopsies of the ectocervix and the endocervix, and assessment for TA treatment. Participants who have a type 1 transformation zone (TZ1) and are otherwise eligible for TA will receive TA with either one or two probes. Screen positive women will be randomized to:

GROUP 1: TA with 1 probe. GROUP 2: TA with 2 probes.

Participants are followed up at 6 months with an HPV test, brush biopsies, and visual assessment of the cervix.

Participants who are not TA eligible will be referred to local care.

ELIGIBILITY:
Inclusion Criteria:

1. 25-49 years old
2. Living with HIV

Inclusion criteria specific to the feasibility study

1. Intact cervix
2. Willing to return to facility at 6 months
3. Willing and able to provide informed consent
4. Positive hrHPV or VIA test within 3 months of enrollment
5. Type 1 transformation zone (TZ1)
6. Thermal ablation eligible

Exclusion Criteria:

1. Screened for cervical cancer outside of study in last 6 months
2. Currently pregnant or less than 6 weeks postpartum
3. Prior diagnosis of cervical cancer
4. A history of treatment for cervical precancer
5. Total hysterectomy
6. Currently receiving treatment for any cancer
7. Individual has a condition that the Clinical Site PI believes will interfere with or affect the conduct, results, or completion of the clinical study
8. Individual has a condition that the Clinical Site PI considers creates an unacceptable risk to the individual if enrolled

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with persistent HPV at 6 months | From enrollment to follow up at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Winer, PhD, MPH, Principal Investigator — University of Washington; Margaret M Madeleine, PhD, MPH, Study Chair — Fred Hutchinson Cancer Center; Leeya Pinder, MD, MPH, Study Chair — University of Cincinnati
Locations (1):
- Research for Development (RD) Rwanda, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
Research data will be shared in a timely manner, with appropriate privacy and confidentiality protections, using the policies and procedures outlined in the NIH Guidelines for Sharing Research Data. Guidelines, oversight, and requirements for sharing data are based on the institutional policies, IRB rules, and local, state, and federal laws and regulations. In all cases, the privacy and confidentiality of all people who participate in the research will be protected. Clinical data on women living with HIV generated during the study will be made available to researchers in both the private and public sector free or for a nominal charge.
Time Frame: Deidentified data, the study protocol, and the data dictionary will be made available to qualified investigators within 6 months of acceptance of the manuscript describing major outcomes, for up to 5 years.
Access Criteria: Requestors will be required to obtain IRB approval and sign a data use agreement before data will be released. The data use agreement must include the following commitments: a commitment to using the data for research purposes only and not to identify any individual participants; a commitment to securing the data using appropriate computer technology; a commitment to destroying or returning the data after analyses are completed; and a commitment to meet any additional requirements that might be stipulated by the RNEC or Fred Hutch regulatory review committees or NCI.